CLINICAL TRIAL: NCT05432011
Title: PENG Block Combined to Lateral Femoral Cutaneous Nerve Block vs. PENG Block Combined to Wound Infiltration for Postoperative Analgesia Following Posterolateral-approached Total Hip Arthroplasty
Brief Title: PENG Block Plus Lateral Femoral Cutaneous Nerve Block for Posterolateral-approached Total Hip Arthroplasty
Acronym: PENG-FLAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Campus Bio-Medico University (Other)
Responsible Party: Principal Investigator, Giuseppe Pascarella, Principal Investigator, Campus Bio-Medico University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PAR 34.22
Record Dates: First submitted 2022-06-20; First posted 2022-06-24 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Pain; Postoperative Pain; Acute Pain; Analgesia; Hip Arthropathy; Postoperative Complications
MeSH Terms: conditions — Pain; Pain, Postoperative; Acute Pain; Agnosia; Postoperative Complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PENG block plus Femoral Cutaneous Nerve Block (Experimental): Participants receiving PENG block combined to Lateral Femoral Cutaneous Nerve Block
  Interventions: Procedure: PENG Block; Procedure: Lateral Femoral Cutaneous Nerve Block
- PENG block plus Wound Infiltration (Active Comparator): Participants receiving PENG block combined to wound infiltration
  Interventions: Procedure: PENG Block; Procedure: Wound Infiltration

INTERVENTIONS:
Procedure: PENG Block — At the end of surgery, in Post Anesthesia Recovery Room (PACU), PENG block with 20 mL of 0.5 % Ropivacaine will be executed as described by Giron-Arango et al. using a low frequency curvilinear probe. A 22G 80 mm needle (Stimuplex Ultra 360, B.Braun) will be used.
Procedure: Lateral Femoral Cutaneous Nerve Block — At the end of surgery, in Post Anesthesia Recovery Room (PACU), ultrasound guided Lateral Femoral Cutaneous Nerve Block will be performed with 10 mL of 0.5 % Ropivacaine using a high frequency linear probe. A 22G 50 mm needle (Stimuplex Ultra 360, B.Braun) will be used.
  Arms: PENG block plus Femoral Cutaneous Nerve Block
Procedure: Wound Infiltration — At the end of operation, the surgeon will perform wound infiltration with 20 mL of 0.5 % Ropivacaine.
  Arms: PENG block plus Wound Infiltration

SUMMARY:
This study aims to analyze the effect of Pericapsular Nerve Group (PENG) Block combined with lateral femoral cutaneous nerve block vs. PENG block combined with wound infiltration for analgesia after elective hip replacement performed with a posters-lateral approach.

Half of participants will receive a PENG Block combined with femoral lateral cutaneous nerve block, while the other half will receive PENG Block combined with wound infiltration

ELIGIBILITY:
Inclusion Criteria:

* Elective hip replacement surgery performed with a poster-lateral approach
* ASA physical status score < 4

Exclusion Criteria:

* Contraindications to regional anesthesia
* ASA physical status score ≥ 4
* Patient's refusal or inability to sign the informed consent
* Allergies to any drug provided by the study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-05-18 (Actual); Study Completion 2023-05-25 (Actual)

PRIMARY OUTCOMES:
Static Pain Score | 24 hours
  A numerical rating scale (NRS) from 0 (no pain) to 10 (worst imaginable pain) will be used to evaluate pain at rest during 24 hours after surgery
Dynamic Pain Score | 24 hours
  A numerical rating scale (NRS) from 0 (no pain) to 10 (worst imaginable pain) will be used to evaluate pain on movement during 24 hours after surgery

SECONDARY OUTCOMES:
Morphine consumption | 24 hours
  Total of intravenous morphine (expressed in milligrams) administered during the first 24 hours after surgery
Morphine consumption | 6 days
  Total of intravenous morphine (expressed in milligrams) administered during the entire hospitalization
Range of hip motion | 24 hours
  Degrees of hip flexion
Quadriceps Strength | 24 hours
  Ability to flex the knee against gravity
Ability to start physiotherapy during the first postoperative day | 24 hours
  YES: the patient was able to start physiotherapy NO: the patient was not able to start physiotherapy during the first postoperative day due to pain or motor block
Ability to ambulate with the help of a walker during the first postoperative day | 24 hours
  YES: The patient was able to ambulate with the help of a walker NO: The patient was not able to ambulate with the help of a walker due to pain or motor block
Incidence of block complications | 24 hours
  Any complications or side effects of the blocks, such as local infection, intravascular injection of local anesthetics and immediate systemic toxicity.
  Moreover, incidence of nausea, vomiting and postoperative respiratory depression will be recorded
Hospital Length of Stay | 6 days
  Total Hospital length of Stay (expressed in days)

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Pascarella, MD, Principal Investigator — University Hospital Campus Biomedico of Rome
Locations (1):
- Campus Bio-medico University Hospital Foundation, Rome, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Pascarella G, Costa F, Del Buono R, Pulitano R, Strumia A, Piliego C, De Quattro E, Cataldo R, Agro FE, Carassiti M; collaborators. Impact of the pericapsular nerve group (PENG) block on postoperative analgesia and functional recovery following total hip arthroplasty: a randomised, observer-masked, controlled trial. Anaesthesia. 2021 Nov;76(11):1492-1498. doi: 10.1111/anae.15536. Epub 2021 Jul 1. PMID 34196965
- [Result] Aliste J, Layera S, Bravo D, Jara A, Munoz G, Barrientos C, Wulf R, Branez J, Finlayson RJ, Tran Q. Randomized comparison between pericapsular nerve group (PENG) block and suprainguinal fascia iliaca block for total hip arthroplasty. Reg Anesth Pain Med. 2021 Oct;46(10):874-878. doi: 10.1136/rapm-2021-102997. Epub 2021 Jul 20. PMID 34290085
- [Result] Giron-Arango L, Peng PWH, Chin KJ, Brull R, Perlas A. Pericapsular Nerve Group (PENG) Block for Hip Fracture. Reg Anesth Pain Med. 2018 Nov;43(8):859-863. doi: 10.1097/AAP.0000000000000847. PMID 30063657
- [Result] Del Buono R, Padua E, Pascarella G, Costa F, Tognu A, Terranova G, Greco F, Fajardo Perez M, Barbara E. Pericapsular nerve group block: an overview. Minerva Anestesiol. 2021 Apr;87(4):458-466. doi: 10.23736/S0375-9393.20.14798-9. Epub 2021 Jan 12. PMID 33432791